CLINICAL TRIAL: NCT02214329
Title: Game-Based Virtual Reality Approach for Improving Balance, Reducing Falls, and Preventing Complications In Diabetes
Brief Title: Sensor-based Balance Training in Diabetes: A Virtual Reality Paradigm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: Qatar National Research Foundation, Qatar (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1100000467
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes
Keywords: Postural Balance; Gait; Fall risk
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensor-based exercise training (Experimental): The intervention group receives sensor-based balance training with real-time joint feedback through an interactive interface on LC monitor screen.
  Interventions: Device: Sensor-based exercise training
- In-home balance training (Active Comparator): The control group performs similar exercise as intervention group at home without use of sensor or any joint feedback from sensor data.
  Interventions: Other: In-home balance training

INTERVENTIONS:
Device: Sensor-based exercise training — Body-worn sensors are mounted on different body segments to acquire joint kinematic data and provide real-time joint feedback during exercise training.
  Arms: Sensor-based exercise training
Other: In-home balance training — The control group performs similar exercise as intervention without sensors and with no visual feedback from sensors.
  Arms: In-home balance training

SUMMARY:
Diabetic peripheral neuropathy (DPN) can severely deteriorate balance and gait in patients, thereby increasing risk of fall and injury. The aim of the study is to evaluate the efficacy of a virtual reality game based exercise training for improving postural body sway and gait in diabetes patients with peripheral neuropathy. The exercise training has been specifically designed for DPN patients with lost lower extremity joint perception and uses state-of-the-art inertial sensors (body-worn) to acquire joint movement and provide real-time joint feedback through an interactive interface on a LCD monitor. The investigators hypothesize that tailored exercise with real-time visual joint feedback during exercise will reduce improve balance and gait.

DETAILED DESCRIPTION:
The game includes a series of ankle reaching tasks and crossing of virtual obstacles on the monitor screen; these exercises are aimed to improve weight shifting capabilities and medial-lateral movement of body.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic peripheral neuropathy
* Age > 50 (Men or Women)
* Able to walk 60 feet

Exclusion Criteria:

* Major lower extremity amputation
* Cognitive deficits (MMSE 24 or below)
* Severely impaired vision

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Postural Balance | 6 weeks
  Postural balance is assess at baseline and post-training using body-worn sensors
Gait | 6 weeks
  Gait is assessed at baseline and post-training using body-worn sensors

SECONDARY OUTCOMES:
Physical Activity | 6 weeks
  Physical activities of daily living are assessed at baseline and post-training using a T-shirt embedded body-worn sensor (PAMSys)
Functional Performance | 6 weeks
  Tests, including 3m timed up and go test and alternative step test, are performed. Time is recorded using a stop watch.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, Tucson, Arizona, United States